CLINICAL TRIAL: NCT06775054
Title: The Role of Cognitive Flexibility in Depression and Response to Transcranial Magnetic Stimulation (TMS)
Brief Title: Cognitive Flexibility in Depression and TMS Response
Acronym: CogFelx_TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Beyazit Garip, Principal Investigator, Gulhane Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-19 / TMS
Record Dates: First submitted 2024-12-29; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Depression - Major Depressive Disorder; Cognitive Flexibility; Treatment Response; Side Effects
Keywords: Depression; TMS; TRD; WCST; TMT; VF
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The Treatment-Resistant Depression (TRD) patient group will be evaluated before and after Transcranial Magnetic Stimulation (TMS) treatment. There will also be a control group consisting of healthy participants, who will undergo a single neuropsychological and clinical assessment. Cognitive flexibility will only be evaluated before the TMS procedure using neuropsychological assessment tools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Flexibility and TMS (Experimental): Treatment resistant depression group Participants will be treated with transcranial magnetic stimulation (TMS) using the MagVenture™ X100™ device. The treatment includes 20 sessions over 4 weeks, delivering 18000 pulses in total. The stimulation targets the left dorsolateral prefrontal cortex, with parameters set to achieve optimal therapeutic effects without inducing adverse side effects. Motor threshold measurements are conducted prior to the initiation of treatment and adjusted weekly to maintain consistent treatment intensity.
  A comprehensive neuropsychological test battery, including the Wisconsin Card Sorting Test (WCST), Trail Making Test (TMT), and Verbal Fluency (VF) tests, was administered to all patients prior to the initiation of treatment. Clinical assessment scales, including the Patient Health Questionnaire-9 (PHQ-9), Clinical Global Impression-Severity (CGI-S), and Clinical Global Impression-Improvement (CGI-I) scales, were administered both before and after TMS
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation (TMS) is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain. It is primarily used to treat depression, particularly in patients who have not responded to traditional treatments such as selective serotonin reuptake inhibitors (SSRIs) or psychotherapy. The most common target area is the dorsolateral prefrontal cortex, which is often underactive in individuals with depression. TMS devices, such as the FDA-approved Magventure system, deliver magnetic pulses to stimulate or inhibit brain activity in the targeted region. This process is believed to help reset or normalize patterns of neural activity associated with depression and other psychiatric disorders. TMS offers a promising alternative for individuals struggling with depression, providing a non-invasive approach with relatively few side effects and notable potential benefits.

SUMMARY:
The primary aim of this study is to determine the level of cognitive flexibility in patients with TRD before treatment and to explore whether there is a relationship with their response to TMS treatment. More specifically, the study aims to identify the role of cognitive flexibility as a neurocognitive marker that could predict whether patients planned to undergo TMS treatment will respond to the treatment. The main focus of this study is to ascertain whether the data obtained have practical implications, particularly regarding the identification of TRD patients who do not respond to TMS treatment in advance.

DETAILED DESCRIPTION:
The primary aim of this prospective study is to determine the level of cognitive flexibility in patients with treatment-resistant depression (TRD) before treatment and to explore whether there is a relationship between cognitive flexibility and their response to TMS treatment. TRD represents a subset of major depressive disorder in which patients do not adequately respond to conventional antidepressant treatments. Emerging evidence suggests that TMS, a noninvasive brain stimulation technique, can effectively alleviate symptoms in TRD patients. However, the Stanford Accelerated Intelligent Neuromodulation Therapy study suggests that 20% of the TRD group may not respond to treatment and could represent an endophenotypic subgroup. In this context, patients with better cognitive flexibility may show a better response to TMS, and the addition of behavioral methods to enhance flexibility could be considered as an adjunct to TMS treatment.

The study will enroll 49 patients diagnosed with treatment-resistant depression (TRD) based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria. Participants will undergo a TMS treatment regimen using the MagVenture™ X100™ device. The treatment protocol will consist of 20 sessions over four weeks, delivering 18,000 pulses in total (using theta burst stimulation). The stimulation will target the left dorsolateral prefrontal cortex, with parameters designed to achieve optimal therapeutic effects while minimizing side effects. Motor threshold measurements will be conducted prior to treatment initiation and adjusted weekly to maintain consistent treatment intensity.

A control group consisting of 65 healthy participants will undergo a single evaluation for neuropsychological and psychometric assessments, with no treatment or follow-up.

Before starting TMS treatment, all patients will undergo a neuropsychological test battery, including the Wisconsin Card Sorting Test (WCST), Trail Making Test (TMT, Verbal Fluency (VF) Tests to determine their cognitive flexibility levels. The Cognitive Flexibility and Control Scale (CFCS), a self-report measure, will be administered to patients who meet the eligibility criteria. Psychiatric assessments will include the Patient Health Questionnaire (PHQ-9) to evaluate changes in depressive symptoms, while the Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) scales will be administered before and after the 20 sessions of TMS treatment.

The primary objective is to assess improvements in symptom severity and the relationship with cognitive flexibility, as measured by the neurocognitive test battery. This will provide valuable insights for clinicians to better understand which patients are most likely to benefit from TMS treatment. The secondary objectives include identifying clinical and neurocognitive features in patients who do not respond to TMS treatment, assessing side effects, and examining whether concurrent medication, such as anti-obsessive medications, influences the efficacy of TMS therapy.This study will offer valuable data for clinicians and researchers, ultimately guiding safer and more effective use of TMS in psychiatric practice.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with Major Depressive Disorder according to DSM-5 TR.

* Diagnosed with Obsessive-Compulsive Disorder according to DSM-5 TR.
* Lack of response to treatment after being administered at least two different antidepressants and anti-obsessive agents at effective doses and durations.
* The clinical condition cannot be better explained by a metabolic or organic disorder.
* Routine electroencephalography (EEG) findings before TMS do not indicate electrical activity consistent with an epileptic focus.
* Routine blood tests before TMS show no conditions that could affect treatment levels, particularly thyroid issues, vitamin deficiencies, or inflammation parameters that might cause depression or cognitive impairment (consultation with relevant departments if necessary).
* No history of hearing loss identified during routine evaluations (if a history of hearing loss exists, consultation will be requested; if none, the process will proceed accordingly).

Exclusion Criteria:

* According to the pre-TMS risk assessment form, there is a contraindication for treatment,
* Epileptic focus is detected in the pre-TMS electroencephalography findings,
* Previous head trauma, loss of consciousness and intra-cerebral surgery,
* A metal particle caused by an aneurysm clip, connection tongs or explosive substances that will affect the electromagnetic field in the brain,
* A significant disorder in the thyroid hormone profile in routine blood checks before TMS,
* A significant increase in inflammation markers in routine checks before TMS,
* A vitamin deficiency that may cause cognitive impairment or forgetfulness in routine blood checks before TMS,
* A presence of electrolyte imbalance in routine blood checks before TMS,
* The patient has previously had a psychotic attack or bipolar mood attack,
* The patient has previously had a substance-induced psychosis or bipolar mood disorder,
* The patient has previously used substances known as alcohol, drugs or stimulants according to DSM-V TR and semi-structured clinical interview (SCID-5 TR) have abuse or addiction (except if they have not used in the last 12 months or have not abused alcohol),
* Those who want to terminate TMS treatment voluntarily, Note:If an unexpected clinical situation occurs during TMS treatment, the patient will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Assessing Cognitive Flexibility in TMS Treatment:WCST | From enrollment to the end of treatment at 4 weeks
  Cognitive flexibility will be evaluated in cases of treatment-resistant depression using a neuropsychological test battery. This battery will be applied only before the TMS treatment.
  Wisconsin Card Sorting Test (WCST): The WCST evaluates cognitive flexibility, problem-solving skills, and executive functioning. It measures an individual's ability to adapt to changing rules or conditions and to shift cognitive strategies when faced with new tasks. This test assesses the ability to overcome perseveration (sticking to an incorrect rule) and adapt to the correct rule based on feedback. The WCST uses a deck of 128 cards, each with one of four shapes (circle, triangle, star, or cross), in one of four colors (red, green, yellow, or blue), and with one of four numbers (1, 2, 3, or 4). It is valuable for understanding how patients adapt to new information, shifting circumstances, and challenges, making it a key part of cognitive evaluations in clinical settings.
Exploring Changes in Task-Switching Ability: The Effect of TMS on TMT Performance | From enrollment to the end of treatment at 4 weeks
  The Trail Making Test (TMT) is a widely used neuropsychological assessment tool designed to evaluate cognitive functions, including executive functioning, cognitive flexibility, visual attention, and processing speed. The test is divided into two parts: TMT-A and TMT-B, each measuring different cognitive aspects.
  Cognitive Aspects Measured by TMT:
  Cognitive Flexibility: The ability to switch between tasks (TMT-B) and adjust strategies is a key indicator of executive functioning. Poor performance on TMT-B may suggest deficits in cognitive flexibility.
  Attention and Processing Speed: TMT-A measures basic processing speed and attention. Delays or errors in completing the test can indicate difficulties with these cognitive domains.
  Executive Functioning: Both parts of the TMT assess aspects of executive functioning, particularly planning, mental flexibility, and working memory.
Evaluating Changes in Verbal Fluency Pre- and Post-TMS Treatment | From enrollment to the end of treatment at 4 weeks
  Verbal fluency (VF) tasks are widely used in neuropsychological assessments to measure cognitive functions such as language production, executive control, and semantic memory. These tasks provide valuable insights into the cognitive abilities of individuals, especially those with psychiatric and neurological conditions. The primary aim of this evaluation is to assess changes in verbal fluency performance in individuals undergoing TMS treatment for depression, specifically treatment-resistant depression. Verbal fluency is commonly assessed through two main types of tasks: Phonemic Fluency: The ability to generate words beginning with a specific letter (e.g., "K" "A," or "S") within a set time limit. Semantic Fluency: The ability to generate words belonging to a specific category (e.g., animals, fruits, etc.) within the same time limit.
Cognitive Flexibility as a Predictor of Transcranial Magnetic Stimulation Outcomes | From enrollment to the end of treatment at 4 weeks
  The relationship between cognitive flexibility, assessed through neuropsychological tests (WCST, TMT, VF), will be evaluated prior to the TMS procedure. For cases of treatment-resistant depression, a ≥ 50% reduction in the PHQ-9 score is generally considered a clinically significant response to treatment. The PHQ-9 score ranges from a minimum of 0, indicating no depressive symptoms, to a maximum of 27, indicating severe depressive symptoms. The interpretation of PHQ-9 scores is as follows: 0-4 indicates minimal or no depression, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Assessing Depression Severity Before and After Transcranial Magnetic Stimulation Treatment | From enrollment to the end of the treatment at 4 weeks.
  A ≥ 50% reduction in the PHQ-9 score is often considered a clinically significant response to treatment. The PHQ-9 scoring ranges from a minimum score of 0, indicating no depressive symptoms, to a maximum score of 27, indicating severe depressive symptoms. The interpretation of PHQ-9 scores is as follows: 0-4 indicates minimal or no depression, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Evaluating Response to TMS Treatment Using the Clinical Global Impression Scale (CGI) | From enrollment to the end of treatment at 4 weeks
  Patients undergoing TMS treatment will be evaluated using the Clinical Global Impression (CGI) scale, which will be applied both before and after the TMS treatment to assess changes in clinical status. The CGI is a standardized tool consisting of two main components: CGI-Severity (CGI-S), which evaluates the severity of the patient's condition on a 7-point scale (1 = normal, 7 = extremely ill), and CGI-Improvement (CGI-I), which assesses the degree of improvement or worsening compared to baseline on a similar 7-point scale (1 = very much improved, 7 = very much worse). This scale provides clinicians with a practical and reliable method for monitoring the effectiveness of treatment and patient progress over time.

SECONDARY OUTCOMES:
Tracking Depression Severity Changes | From enrollment to the end of treatment at 4 weeks
  Depressive symptoms will be evaluated using the Patient Health Questionnaire (PHQ-9) both before and after the TMS treatment to assess the effectiveness of the TMS protocol. The PHQ-9 is a widely used self-administered tool consisting of nine questions designed to assess the severity of depression symptoms experienced over the past two weeks. Each question is rated on a scale from 0 to 3, where 0 indicates no symptom and 3 represents the most severe symptom. The total score, which ranges from 0 to 27, provides a quantitative measure of depressive symptom severity. Higher scores on the PHQ-9 indicate more intense depressive symptoms.
  For the purpose of evaluating treatment response, a greater than 50% reduction in the PHQ-9 score following the TMS treatment will be considered indicative of a positive response to the therapy. This significant reduction in score reflects a marked improvement in depressive symptoms, signaling the effectiveness of the TMS protocol.
Side Effect Assessment | From enrollment to the end of treatment at 4 weeks
  Recording any adverse events or unexpected side effects noted during or after the transcranial magnetic stimulation (TMS) sessions, to evaluate the safety profile of the treatment. There is no standardized method for evaluating the side effects of TMS, a clinician will evaluate the participants for known side effects including changes in hearing, local pain, muscle contractions, headache, non-specific tingling, and discomfort.
Drug Interaction Effects | From enrollment to the end of treatment at 4 weeks
  Drug interactions during TMS treatment will be assessed using the TMS side effect questionnaire. Medications that lower the seizure threshold, such as bupropion, will be documented prior to the TMS procedure. During the procedure, any side effects, such as headaches and intense application site pain, will be evaluated using the Visual Analog Scale (VAS). The Visual Analog Scale (VAS) consists of a straight line, typically 10 cm long (or sometimes 100 mm), where one end represents no symptoms (e.g., "0" or "no pain") and the other end represents the most severe symptoms imaginable (e.g., "10" or "worst possible pain"). Patients are asked to mark a point on the line that corresponds to the severity of their symptom, and this point is then measured in centimeters or millimeters to provide a numerical score reflecting the intensity of the symptom. The minimum value (0) represents no symptoms at all, such as "no pain" or "no nausea," while the maximum value (10) represents the most intense

CONTACTS AND LOCATIONS:
Overall Officials: BEYAZIT GARİP, Medical Doctor, Principal Investigator — Gulhane Trainin and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IDP) will be shared together with the Clinical Study Report
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be made available immediately after the publication, and will remain available for at least 5 years.
Access Criteria: Anyone who wishes to access the data